CLINICAL TRIAL: NCT03424668
Title: The European Prospective Investigation Into Cancer in Norfolk Prospective Population Study
Acronym: EPIC-Norfolk
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Medical Research Council (Other Government); Cancer Research UK (Other)
Responsible Party: Principal Investigator, Kay-Tee Khaw, Professor of Clinical Gerontology, University of Cambridge
Other Study IDs: MR/N003284/1
Record Dates: First submitted 2018-01-25; First posted 2018-02-07 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Neoplasms; Cardiovascular Diseases; Death
Keywords: nutrition; physical activity; lifestyle; smoking
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Death; Motor Activity; Smoking | interventions — Diet; Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: diet — lifestyle factors
  Other Names: physical activity

SUMMARY:
The European Prospective Investigation into Cancer and Nutrition in Norfolk is a population based prospective study of approximately 25,000 men and women resident in Norfolk United Kingdom. They were aged 39-79 years when first recruited from general practice age sex registers at baseline assessment 1993-1997. While part of a ten country half million participant European collaboration originally aimed to investigate diet and other lifestyle determinants of cancer, the objectives of the Norfolk cohort from inception were expanded to encompass the trajectory of health, ill health and mortality in a population over time and to examine the biological and lifestyle determinants of health and chronic disease.

DETAILED DESCRIPTION:
The European Prospective Investigation into Cancer and Nutrition in Norfolk is a population based prospective study of approximately 25,000 men and women resident in Norfolk United Kingdom. They were aged 39-79 years when first recruited from general practice age sex registers at baseline assessment 1993-1997. While part of a ten country half million participant European collaboration originally aimed to investigate diet and other lifestyle determinants of cancer, the objectives of the Norfolk cohort from inception were expanded to encompass the trajectory of health, ill health and mortality in a population over time and to examine the biological and lifestyle determinants of health and chronic disease. Detailed data on sociodemographic, lifestyle, medical and family history were collected and a biological sample bank including urine and blood samples established. Participants have been followed up through repeat examinations, mailed questionnaires as well as through record linkage with routine health records including death certification by cause, cancer registration and hospital admissions by cause till present.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* On general practice age sex registers in Norfolk, United Kingdom in 1993-1997

Exclusion Criteria:

* Not willing to participate in study
* terminal illness

Ages: 39 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Resident in Norfolk, United Kingdom on general practice age sex registers 1993-1997
Sampling Method: Non-Probability Sample
Enrollment: 25639 (Actual)
Dates: Start 1992-01-01 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
neoplasms | Through 25 years
  cancer incidence

SECONDARY OUTCOMES:
cardiovascular diseases | through 25 years
  incidence of cardiovascular diseases
death | through 25 years
  total mortality by cause

OTHER OUTCOMES:
fractures | through 25 years
  incident fractures
diabetes mellitus | through 25 years
  incident diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Wareham, MBBS, Principal Investigator — University of Cambridge; Kay-Tee Khaw, MBBChir, Principal Investigator — University of Cambridge

IPD SHARING:
Plan to Share IPD: Yes
EPIC Norfolk follows Medical Research Council UK good practice for data sharing. Requests for data are submitted to the EPIC Norfolk management committee to assess scientific feasibility and avoid duplication and within the requirements of NHS Digital data protection rules.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data are available after collection, cleaning and quality control
Access Criteria: Bonafide researchers
URL: http://www.srl.cam.ac.uk/epic/

REFERENCES:
- [Background] Day N, Oakes S, Luben R, Khaw KT, Bingham S, Welch A, Wareham N. EPIC-Norfolk: study design and characteristics of the cohort. European Prospective Investigation of Cancer. Br J Cancer. 1999 Jul;80 Suppl 1:95-103. No abstract available. PMID 10466767
- [Background] Bingham SA, Welch AA, McTaggart A, Mulligan AA, Runswick SA, Luben R, Oakes S, Khaw KT, Wareham N, Day NE. Nutritional methods in the European Prospective Investigation of Cancer in Norfolk. Public Health Nutr. 2001 Jun;4(3):847-58. doi: 10.1079/phn2000102. PMID 11415493